CLINICAL TRIAL: NCT02884193
Title: Effects of Brief and Prolonged Cold Application on Maximal Isometric Hand Grip Strength.
Brief Title: Cold and Isometric Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Principal Investigator and Clinical Professor, Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6031206
Record Dates: First submitted 2016-08-10; First posted 2016-08-30 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-02

CONDITIONS: Muscle Strength
Keywords: Cooling; Cryotherapy; isometric Strength; Palmar Grip; Dynamometry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Cooling (Quick Icing) (Experimental): Group receiving the application of cold on the ventral side of the dominant forearm for 30 seconds, using the technique of ice beakers dynamically.
  Interventions: Procedure: Brief Cooling
- Prolonged Cold (Active Comparator): Group receiving the intervention of "ice bag" for a period of 5 and a half minutes from 1 minute, on the ventral side of the dominant forearm
  Interventions: Procedure: Prolonged Cold
- Control (Sham Comparator): Group receives a placebo application through an "ice bag" empty. The bag will be applied from 1 minute to 6 and a half minutes, as the group of prolonged cold
  Interventions: Procedure: Sham Ice Bag

INTERVENTIONS:
Procedure: Brief Cooling — Brief Application of cold, for a period of up to 30 seconds on a body surface which seeks to promote the activation of the nervous system to produce increased excitability.
  Other Names: Quick Icing
  Arms: Brief Cooling (Quick Icing)
Procedure: Prolonged Cold — Prolonged application of cold, for at least 5 minutes or more, on a body surface that aims to reduce nervous system activation by reducing the NCV.
  Arms: Prolonged Cold
Procedure: Sham Ice Bag — Placebo application through an "ice bag" empty.
  Arms: Control

SUMMARY:
Cryotherapy has a wide range of clinical applications in rehabilitation, used for activities such as controlling inflammation, pain control or management of edema after an injury or surgery. In the field of cryotherapy they studied cold neuromuscular responses, where it has shown a decrease in nerve conduction velocity, which leads to a decrease in muscle strength. However it has been described in some work applications brief cold ("Quick Icing") may be opposite to those described effects, increasing the strength, the time of intervention the most important and decisive in these possible improvements or decreases factor. This effect is observed in response to a few seconds of application of cold, and would be given by an increased activity of motor neurons. Assess the influence of rapid cooling application ("Technique Quick Icing") and prolonged cooling in handgrip strength when performing a manual dynamometer test in college students.

DETAILED DESCRIPTION:
Methodology

1. Type of study: Experimental study, type randomized clinical trial (RCT).
2. Conceptual framework:

   * Quick or rapid cooling Icing: brief application of cold, for a period of up to 30 seconds on a body surface which seeks to promote the activation of the nervous system to produce increased excitability.
   * Prolonged Cold: prolonged application of cold, for at least 5 minutes or more, on a body surface that aims to reduce nervous system activation slowing of nerve conduction.
3. Operational definition of variables:

   * Grip strength: Strength in kilograms evaluated through manual dynamometry test the time for a grip. Force values are recorded in an Excel table displaying data in kilograms evaluated. (Manual hydraulic dynamometer brand JAMAR® be used).
   * Quick Icing: will apply through glasses of ice on the ventral region of the dominant forearm of the experimental group.
   * Prolonged cold: It shall be implemented through an ice pack (ice bag), placed on the ventral side of the dominant forearm in one of the comparison groups.
   * Control: Group of people will not be subjected to any intervention.
4. Sample:

   Place of research: The study will be conducted in the laboratory of physiotherapy rehabilitation science faculty building C5 401 room floor room, campus Casona de la Universidad Andrés Bello, Av Fernández Concha 700, Las Condes.
5. Methodological Design

This research has the characteristics of a random analytical experimental design (ECA), the study will be conducted in the laboratory Intervention Kinesics, room 401, fourth floor C5, Faculty of Rehabilitation Sciences, Campus Casona Las Condes, Av. Fernández Concha 700, Comuna Las Condes. The sample will be selected from the university community that makes up the faculty of Rehabilitation Sciences (FCR). The research will be registered in the network of clinical trials registry (www.clinicaltrials.gov), obtaining a registration number. The study has submitted to the ethics committee of the East Metropolitan Health Service (SSMO), to ensure that all bioethical labor standards are met. It is approved on August 23, 2016. This allowed to start the investigation. Population will be taken as students who are studying between first and fourth year of racing Kinesiology, Speech Therapy and Occupational Therapy. The sample is determined by a deliberate selection process through a survey of closed questions. This survey will allow participants to choose from the selection criteria proposed in the work. The number of participants that make up the sample will be taken for the convenience of researchers. As inclusion criteria have been established which follow: Students of the Faculty of Rehabilitation Sciences UNAB, subjects older than 18 years and have not submitted musculoskeletal disorders in the dominant upper extremity in the last 6 months. Moreover, as exclusion criteria have been considered: the presence of pain or discomfort in performing handgrip with the dominant limb, intolerance to cold, diseases such as cryoglobulinemia, Raynaud's disease or paroxysmal hemoglobinuria cold, rheumatic diseases such as lupus erythematosus systemic, multiple myeloma or rheumatoid arthritis, positive test cube ice and osteosynthesis materials or stent in the dominant upper extremity. The exclusion criteria will be assessed in the sampling process through the selection of survey participants.

They have designated three stages of conducting the study. Stage 1, called "Stage sampling" consist of the application of the survey to students of different levels of the three races of the faculty. Then it analyzes information collected by performing a first filter in selecting potential participants. This filter is given by the survey questions that reflect the inclusive and exclusive criteria. Personal contact with students who meet the characteristics of participation and will be invited to join the study will be conducted. A selectable and interested in participating they will be explained the purpose of the investigation and asked for their consent to participate in writing. The document will be given consent previously approved by the bioethics committee of the East Metropolitan Health Service (SSMO), based in the Salvador Hospital, Providence commune. Stage 1 will be as lasting three weeks, following the planned proposal on the Gantt chart.

The second stage of the design, called "Evaluation" will last for two weeks according to the proposal in the Gantt chart established. This step will be the completion of the ice cube test following the established protocol. This will apply a second filter of selectable subjects and who agreed to participate consentidamente, and not excluded from the survey team. Then an assessment of the ability of participants will be made to perform painless handgrip on a stage with the same environmental conditions in which they carry out research (laboratory Physiotherapy Faculty Rehabilitation Sciences, Room 307, fourth floor building C5 ). Thus the stage 2 will be an instance of second filtering selection of participants, to have people who eventually will make up the working groups of the study.

Stage 3, called "Experimental", will run for eight weeks. Participants will be distributed forming three working groups, a group called "Quick Icing" (QI), another group called "Prolonged Cold" (PC) and a third group called "Control" (C). The designation for each group will advance by a simple randomization process using a table of random numbers, and will be in charge of the study director. Thus each participant will be labeled with a number and included in a specific group. This randomization process will seek to minimize selection bias. The director will be the only one who has the numbered list of participants in each group. From this process of randomization working groups will be established, that is, "Quick Icing", "Prolonged cold" and "Control". After forming the three groups, an evaluator 1 record demographic characteristics of each participant. This record will include data such as; age, body mass index (BMI), gender and body fat percentage. This information will be extracted from the survey participant selection that will form groups and measuring the percentage of body fat.

In analysis of these data will determine the homogeneity of the groups to establish any comparisons at the end of the process after having results. An evaluator 2, unknown belongs to each participant, record the maximum handgrip strength of the dominant limb of each individual. The maximum handgrip strength will be evaluated following the proposed design the test protocol using manual dynamometry, registering the force of subjects measured in kilograms (kg). The evaluator 2 shall request three executions within a period of 15 seconds leaving a rest interval of 60 seconds between each attempt, this according to the protocol proposed by the researchers, based on the work of Watanabe and cols.

The evaluator 2 tabulate the values of the three executions in an Excel spreadsheet marking the mean handgrip strength valoe will be recorded as the "pre" maximum force. Followed by the assessment process handgrip strength, we will lead each participant to the intervention group that corresponds, ie group "Quick icing" group "Prolonged Cold" or "Control". In the laboratory has established three working box, one for each intervention procedure. People will only have contact with subjects pertaining to your workgroup, without knowing participants in the other groups, this will be achieved with the double-blind establish avoiding bias intervention. Each participant will be seven minutes in their respective work box. The first minute of the time in question is used for the installation of each individual, leaving the remaining 6 for the application of the procedure. The protocol will consist of installation position the person seated, supporting the dominant forearm on a table leaving visible the ventral side of the segment. The participants of the group "Quick icing" will be subject to the application of cold on the ventral side of the dominant forearm for 30 seconds, using the technique of ice beakers dynamically. Participants must wait in the box six minutes before the therapeutic intervention. The quick icing process will be applied from 6 minutes for the time described above. The group of "prolonged Cold" will receive the intervention of "ice bag" for a period of 5 and a half minutes from 1 minute on the ventral side of the dominant forearm. The "Ice Bag" will have a weight of 700 grams. The "Control" group will receive a placebo application through an "ice bag" empty. The bag will be applied from 1 minute to 6 and a half minutes, as prolonged cold group. After 7 minutes of individuals in each group will return to the station where the evaluator 2 dynamometry record the handgrip strength of the dominant segment in your Excel spreadsheet tabulating the best record of three possible attempts again. This will get the value of maximum force "post" of people in each group.

He completed the "experimental stage" proceed to step 4 called "Data Analysis" which will last for three weeks to allow the ordering of data, development of descriptive and inferential statistics. This stage will lead the research director, who will be responsible for storing and organizing data collected by the evaluators. Descriptive statistics for the variable maximum isometric muscle strength pre and post, will be from intragroup and intergroup averages. Secondary variables age and body mass index will be described in terms of average and standard deviation. The secondary endpoint genre will be described in terms of frequencies and percentages. To represent the descriptive statistics of the variable maximum force, graphic boxes, which show the averages will be used. For each variable statistical Kruskal-Wallis one-way analysis of variance was applied to determine the normal distribution of the data, and thus assess whether there are significant differences in these parameters. To make this analysis STATA ® program will be used. According to normal or abnormal distribution data obtained ANOVA statistical test or SHARIPO-WILK be used. The results from these statistical tests allow the preparation of Table 1 (demographic data), which will reflect the initial data of the participants in each group. Following the framework of inferential statistics will proceed to compare differences in mean maximal isometric forces pre- and post intragroup and intergroup using ANOVA statistical test or Kruskal-Wallis depending on whether the distribution of these variables was normal or abnormal. The analysis will also consider the differences in the mean values of maximum force considering the variable intra- and inter-group genre. Once the statistical analysis done, it is considered two weeks to analyze the results and approach a discussion around them.

After completed all stages of design, we will proceed to spread the work through the application to national and international scientific journals, it will be drafted in accordance with the regulations required by the journal to which it will run. It has seen a period of three months for the dissemination of research.

Parallel each stage of the design will be registered on the clinicaltrials.gov mode page report the status of the investigation.

7. Procedures

Ice Cube Test

1. Subject seated.
2. Shoulder adducted without rotation.
3. Elbow flexed at 90 °. This is ensured by a splint.
4. Forearm in supination.
5. Placing an ice cube on the ventral side of the contralateral forearm during a time of 5 minutes.
6. Unwanted response like hives, blisters, cold intolerance, severe erythema or pain is observed.

Palmar Grasping Protocol

1. Subject seated.
2. Shoulder adducted without rotation.
3. Elbow flexed at 90 °. This is ensured by a splint.
4. Forearm supination neutral Prone.
5. Wrist in a neutral position, that is, spread between 0 and 30, with ulnar deviation from 0 to 15 degrees.
6. Gripping palmar in 3 attempts, recording the best value of maximum force obtained when performing the maneuver.
7. Standing Time 60 seconds between each attempt, this recovery the muscle ATP.

ELIGIBILITY:
Inclusion Criteria:

* Students of the Faculty of Rehabilitation Sciences University Andres Bello.
* Over 18 years.
* No skeletal muscle pathologies of the dominant upper extremity in the last 6 months.

Exclusion Criteria:

* Presence of pain or discomfort in the grip.
* Cold intolerance.
* Pathologies as cryoglobulinemia, Raynaud's disease or paroxysmal cold hemoglobinuria.
* Rheumatoid diseases such as systemic lupus erythematosus, multiple myeloma or arthritis Reumtoide.
* Adverse ice cube test (test positive) reactions.
* Osteosynthesis materials or stent in the dominant upper limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Comparing maximum grip strength pre and post application of cold. | Baseline and 2 hours later (1 session of treatment)
  Force in kilograms evaluated through manual dynamometry test the time for a grip.

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Andrés de la Barra Ortiz, Mg, Principal Investigator — Universidad Andrés Bello
Locations (1):
- Universidad Andrés Bello, Santiago, Comuna Las Condes, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewis M, Clayfield J. Temperature changes following quick icing: a brief investigation. Aust J Physiother. 1981 Dec;27(6):175-8. doi: 10.1016/S0004-9514(14)60756-X. PMID 25025468
- [Background] Watanabe T, Owashi K, Kanauchi Y, Mura N, Takahara M, Ogino T. The short-term reliability of grip strength measurement and the effects of posture and grip span. J Hand Surg Am. 2005 May;30(3):603-9. doi: 10.1016/j.jhsa.2004.12.007. PMID 15925174
- [Background] O'Driscoll SW, Horii E, Ness R, Cahalan TD, Richards RR, An KN. The relationship between wrist position, grasp size, and grip strength. J Hand Surg Am. 1992 Jan;17(1):169-77. doi: 10.1016/0363-5023(92)90136-d. PMID 1538102
- [Background] Boyer J, Fraser J, Doyle A. The hemodynamic effect of cold inmersion, Clin Sci 19:539-543, 1980.
- [Background] Goff B. The application of recent advances in neurophysiology to Miss M. Rood's concept of neuromuscular facilitation. Physiotherapy. 1972 Dec 10;58(12):409-15. No abstract available. PMID 4668364
- [Background] Krumhansl BR. Ice lollies for ice massage. Phys Ther. 1969 Oct;49(10):1098. doi: 10.1093/ptj/49.10.1098. No abstract available. PMID 5343549
- [Background] Knutsson E. Topical cryotherapy in spasticity. Scand J Rehabil Med. 1970;2(4):159-63. No abstract available. PMID 5523762
- [Background] Oliver RA, Johnson DJ, Wheelhouse WW, Griffin PP. Isometric muscle contraction response during recovery from reduced intramuscular temperature. Arch Phys Med Rehabil. 1979 Mar;60(3):126-9. PMID 485802
- [Background] Lee JM, Warren MP, Mason SM. Effects of ice on nerve conduction velocity. Physiotherapy. 1978 Jan;64(1):2-6. No abstract available. PMID 628689
- [Background] CLARKE RS, HELLON RF, LIND AR. Vascular reactions of the human forearm to cold. Clin Sci. 1958 Feb;17(1):165-79. No abstract available. PMID 13511729
- [Background] McGown HL. Effects of cold application on maximal isometric contraction. Phys Ther. 1967 Mar;47(3):185-92. doi: 10.1093/ptj/47.3.185. No abstract available. PMID 6042350
- [Background] Belitsky RB, Odam SJ, Hubley-Kozey C. Evaluation of the effectiveness of wet ice, dry ice, and cryogenic packs in reducing skin temperature. Phys Ther. 1987 Jul;67(7):1080-4. doi: 10.1093/ptj/67.7.1080. PMID 3602101
- [Background] Chesterton LS, Foster NE, Ross L. Skin temperature response to cryotherapy. Arch Phys Med Rehabil. 2002 Apr;83(4):543-9. doi: 10.1053/apmr.2002.30926. PMID 11932859